CLINICAL TRIAL: NCT04466423
Title: Intervention Trial Designed to Promote Collegiality and Mutual Support at Work as a Way to Increase Meaning in Work and Reduce Burnout
Brief Title: Intervention Trial to Increase Meaning in Work and Reduce Burnout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Colin West, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-004834
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Burnout, Professional
Keywords: well-being; burnout
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Groups labeled "1" or "2" with random order assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small group intervention (Experimental): Those randomized to the immediate intervention arm will be asked to meet approximately every other week for 6 months, covering 12 sessions. We will ask each group to meet in a relatively private setting (e.g., a restaurant near campus or a reserved meeting room), rather than more public spaces (e.g. river room, cafeteria) where interruptions are more likely.
  Interventions: Behavioral: Small group meetings (COMPASS: COlleagues Meeting to Promote And Sustain Satisfaction)
- Control (Placebo Comparator): Participants randomized to Arm 2 (delayed intervention) will be "wait listed" to begin sessions 6 months after the start of the study. This participation will be optional.
  Interventions: Behavioral: Small group meetings (COMPASS: COlleagues Meeting to Promote And Sustain Satisfaction)

INTERVENTIONS:
Behavioral: Small group meetings (COMPASS: COlleagues Meeting to Promote And Sustain Satisfaction) — The first 15 minutes of each session will be semi-structured discussion involving i) check in and ii) dialogue about the assigned question. Group leaders will be provided 3-4 discussion questions for each session. The group (or the leader) can choose the one they are most interested in and will then spend 10-15 minutes discussing the question together. Questions will touch on key themes for discussion (see the attached topics list) and are derived from our previous intervention studies. The remainder of the time can be used for socializing and building relationships with colleagues.

SUMMARY:
Collegiality is a one of the great virtues of physician-hood. Mutual support from colleagues to help deal with the challenges of being a physician has long helped physicians manage the stress related to practicing medicine and helped physicians derive meaning from their work. Unfortunately, increased productivity expectations and other changes to the practice of medicine over the last several decades have decreased the time physicians have to interact with colleagues and eroded the fabric of collegiality. Recent studies suggest burnout affects nearly half of U.S. physicians at any given point in time and has substantial personal and professional consequences. The steps organizations can take to promote collegiality are unknown. The goal of the present study is to evaluate the ability of an organizational intervention to encourage collegiality, shared experience, connectedness, and mutual support. This study builds on two prior intervention studies directed by the Mayo Clinic Department of Medicine Program on Physician Well-Being, the first focusing on a small group facilitated well-being curriculum and the second focusing on individual electronic tasks to prompt positive reflection and gratitude.

ELIGIBILITY:
Inclusion Criteria:

* Senior Associate Consultants and Consultants in the Mayo Clinic Department of Medicine will be eligible for this study.

Exclusion Criteria:

* None beyond inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2014-10-01 (Actual)

PRIMARY OUTCOMES:
Burnout | 12 month outcomes
  Maslach Burnout Inventory results

SECONDARY OUTCOMES:
Depressive symptoms | 12 month outcomes
  PRIME-MD
Quality of life | 12 month outcomes
  LASA QOL
Job satisfaction | 12 month outcomes
  PJSS
Meaning at work | 12 month outcomes
  EWS
Social support | 12 month outcomes
  Social Provisions Scale
Social isolation | 12 month outcomes
  PROMIS Social Isolation
Job turnover | 12 month outcomes
  Single item asking about 2-year plans to leave current practice

CONTACTS AND LOCATIONS:
Overall Officials: Colin West, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] West CP, Dyrbye LN, Satele DV, Shanafelt TD. Colleagues Meeting to Promote and Sustain Satisfaction (COMPASS) Groups for Physician Well-Being: A Randomized Clinical Trial. Mayo Clin Proc. 2021 Oct;96(10):2606-2614. doi: 10.1016/j.mayocp.2021.02.028. Epub 2021 Aug 5. PMID 34366134
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials